CLINICAL TRIAL: NCT00576069
Title: Evaluation of Mechanism(s)Limiting Expiratory Airflow in Chronic, Stable Asthmatics Who Are Non-smokers
Brief Title: Mechanism(s)of Airflow Limitation in Moderate-severe Persistent Asthma
Status: Recruiting | Type: Observational
Sponsor: Gelb, Arthur F., M.D. (Individual)
Responsible Party: Principal Investigator, Arthur F Gelb MD, Principal Investigator, Gelb, Arthur F., M.D.
Other Study IDs: 20070934
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Asthma
Keywords: asthma; lung function; inflammation
MeSH Terms: conditions — Asthma; Inflammation | interventions — Budesonide, Formoterol Fumarate Drug Combination; Formoterol Fumarate; Fluticasone-Salmeterol Drug Combination; Mometasone Furoate; Mometasone Furoate, Formoterol Fumarate Drug Combination; Prednisone; Methylprednisolone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- asthma, quality of life, lung function: All Asthmatics will be treated with 1 of 3 long acting beta 2 agonist + corticosteroid using low or medium dose of inhaled (Advair) fluticasone or equivalent corticosteroid 200-500mcg/day plus salmeterol 100 mcg/day or (Symbicort) budesonide 320-640 mcg +formoterol 18 mcg/day or (Dulera) mometasone 400-800mcg + formoterol 20 mcg/day. In addition tiotropium 18ucg/day will be used. Additionally, albuterol 0.083%/ipratropium 0.02% solution or MDI HFA for acute exacerbation.Will measure lung function and asthma quality of life questionaire
  Interventions: Drug: budesonide/formoterol; Drug: fluticasone/salmeterol; Drug: mometasone/formoterol; Drug: Prednisone

INTERVENTIONS:
Drug: budesonide/formoterol — 2 inhalations 2X/daily in treated arm/group. No placebo group
  Other Names: symbicort 80/4.5; symbicort 160/4.5; budesonide 80 or 160ug/formoterol 4.5ug, 2 inhalations bid; spiriva handihaler or respihaler
Drug: fluticasone/salmeterol — fluticasone 100ug/salmeterol 50ug, 1 inhalation bid noplacebo fluticasone 250ug/salmeterol 50ug, 1 inhalations bid no placebo Spiriva handihaler daily or respihaler 2 inhalations daily no placebo group
  Other Names: advair 100/50; advair 250/50
Drug: mometasone/formoterol — 200/5 mcg two puffs bid 100/5 mcg two puffs bid Breo Ellipta once daily Spiriva capsule handihaler once daily or Spiriva respihaler 2 in
  no placebo group
  Other Names: Dulera
Drug: Prednisone — 0-15 mg daily as needed
  Other Names: medrol

SUMMARY:
The purpose of this study is to evaluate the site and mechanisms responsible for expiratory airflow limitation in chronic, treated, non-smoking, stable asthmatics with moderate to severe persistent expiratory airflow obstruction. Treatment will include inhaled corticosteroids and long acting beta2agonists and long acting muscarinic antagonists. We are interested in determining whether the large and/or small airways are the predominant site of airflow limitation. We are also interested in determining whether intrinsic small airways obstruction and/or loss of lung elastic recoil is responsible for expiratory airflow limitation and to what extent may be attributed to loss of lung elastic recoil vs decreased airway conductance in peripheral airways. We are also interested to evaluate the role of varying doses of inhaled corticosteroids to suppress large and small airway inflammation using exhaled nitric oxide as surrogate markers of inflammation. For comparison purposes, spirometry and measurements of exhaled nitric oxide will also be obtained if possible during a naturally occurring exacerbation of asthma. High resolution thin section CT of the lung will also be obtained. Analysis will evaluate integrity of the lung parenchyma as to absence and or presence of emphysema and extent of emphysema using voxel quantification. We will also investigate optical coherence tomography to detect clinically unsuspected emphysema. We will also obtain autopsy material when available in asthmatics who expire. Will also measure serum periostin as a marker of inflammation by collaborating with Genetech in San Francisco.

DETAILED DESCRIPTION:
Results will be evaluated during exacerbation and when stable following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Current non-smoking (<10 pack yr smoking history)
* Stable, treated asthmatics
* Age 12-95 yr
* post 180ug albuterol by MDI: FEV 1/FVC < 70% and FEV 1 <80% predicted

Exclusion Criteria:

* Pregnancy

Ages: 10 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic Asthmatics
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-10-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
use exhaled nitric oxide as a surrogate marker of large airway vs small airway/lung inflammation following various doses of inhaled corticosteroids | 20-60 days
determine site of airflow limitation, whether predominantly large and /or small airways using expiratory flow volume curves obtained before and after asthmatics breathe a 80% helium-20% oxygen gas mixture | 20-60 days
investigate the mechanisms that limit expiratory airflow: intrinsic airway obstruction vs loss of lung elastic recoil | 20-60 days
determine the extent of asthma and distribution of emphysema | within 10 days following death or explanted lung if lung transplant obtained
  at autopsy or post lung transplantation

SECONDARY OUTCOMES:
dynamic hyperinflation | 20-60 days
Evaluate large and small airways and lung parenchyma in autopsied or transplanted lung in asthmatics and look for unsuspected emphysema | June 2018
  If approved by surviving power of attorney, chronic non-smoking asthmatics who expire will undergo autopsy evaluation to evaluate extent of airway obstruction as well as presence of emphysema
Optical Coherence Tomography | June 2015
  When stable, chronic non-smoking asthmatics with persistent expiratory airflow obstruction will undergo OCT via flexible bronchoscopy to detect unsuspected emphysema.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur F Gelb, MD, Principal Investigator — Arthur F Gelb Medical Corporation
Locations (1):
- Arthur F Gelb Medical Corporation, Lakewood, California, United States

IPD SHARING:
Plan to Share IPD: Yes
see publications

REFERENCES:
- [Background] Gelb AF, Zamel N. Unsuspected pseudophysiologic emphysema in chronic persistent asthma. Am J Respir Crit Care Med. 2000 Nov;162(5):1778-82. doi: 10.1164/ajrccm.162.5.2001037. PMID 11069812
- [Background] Gelb AF, Licuanan J, Shinar CM, Zamel N. Unsuspected loss of lung elastic recoil in chronic persistent asthma. Chest. 2002 Mar;121(3):715-21. doi: 10.1378/chest.121.3.715. PMID 11888951
- [Background] Gelb AF, Gutierrez CA, Weisman IM, Newsom R, Taylor CF, Zamel N. Simplified detection of dynamic hyperinflation. Chest. 2004 Dec;126(6):1855-60. doi: 10.1378/chest.126.6.1855. PMID 15596684
- [Background] Gelb AF, Flynn Taylor C, Shinar CM, Gutierrez C, Zamel N. Role of spirometry and exhaled nitric oxide to predict exacerbations in treated asthmatics. Chest. 2006 Jun;129(6):1492-9. doi: 10.1378/chest.129.6.1492. PMID 16778266
- [Background] Gelb AF, Taylor CF, Nussbaum E, Gutierrez C, Schein A, Shinar CM, Schein MJ, Epstein JD, Zamel N. Alveolar and airway sites of nitric oxide inflammation in treated asthma. Am J Respir Crit Care Med. 2004 Oct 1;170(7):737-41. doi: 10.1164/rccm.200403-408OC. Epub 2004 Jun 30. PMID 15229098
- [Background] Gelb AF, Zamel N, Krishnan A. Physiologic similarities and differences between asthma and chronic obstructive pulmonary disease. Curr Opin Pulm Med. 2008 Jan;14(1):24-30. doi: 10.1097/MCP.0b013e3282f197df. PMID 18043272
- [Result] Gelb AF, Moridzadeh R, Singh DH, Fraser C, George SC. In moderate-to-severe asthma patients monitoring exhaled nitric oxide during exacerbation is not a good predictor of spirometric response to oral corticosteroid. J Allergy Clin Immunol. 2012 Jun;129(6):1491-8. doi: 10.1016/j.jaci.2012.03.036. Epub 2012 May 2. PMID 22560478
- [Result] Gelb AF, Yamamoto A, Mauad T, Kollin J, Schein MJ, Nadel JA. Unsuspected mild emphysema in nonsmoking patients with chronic asthma with persistent airway obstruction. J Allergy Clin Immunol. 2014 Jan;133(1):263-5.e1-3. doi: 10.1016/j.jaci.2013.09.045. Epub 2013 Nov 28. No abstract available. PMID 24290280
- [Result] Gelb AF, Singh DH, Moridzadeh R, Fraser C, Tran D, Verbanck S, George SC. Age-stratified comparison of large and peripheral airway/alveolar nitric oxide levels in children and young adults. J Allergy Clin Immunol. 2013 Nov;132(5):1222-4. doi: 10.1016/j.jaci.2013.05.045. Epub 2013 Aug 6. No abstract available. PMID 23932460
- [Result] Gelb AF, Yamamoto A, Verbeken EK, Nadel JA. Unraveling the Pathophysiology of the Asthma-COPD Overlap Syndrome: Unsuspected Mild Centrilobular Emphysema Is Responsible for Loss of Lung Elastic Recoil in Never Smokers With Asthma With Persistent Expiratory Airflow Limitation. Chest. 2015 Aug;148(2):313-320. doi: 10.1378/chest.14-2483. PMID 25950858
- [Result] Gelb AF, Nadel JA. Understanding the pathophysiology of the asthma-chronic obstructive pulmonary disease overlap syndrome. J Allergy Clin Immunol. 2015 Sep;136(3):553-5. doi: 10.1016/j.jaci.2015.06.013. No abstract available. PMID 26343939
- [Result] Gelb AF, Christenson SA, Nadel JA. Understanding the pathophysiology of the asthma-chronic obstructive pulmonary disease overlap syndrome. Curr Opin Pulm Med. 2016 Mar;22(2):100-5. doi: 10.1097/MCP.0000000000000236. PMID 26717511
- [Derived] Gelb AF, Yamamoto A, Verbeken E, Grigorian SR, Nadel JA. Asthma and emphysema overlap in nonsmokers. Ann Allergy Asthma Immunol. 2020 Dec;125(6):711-713. doi: 10.1016/j.anai.2020.08.010. Epub 2020 Aug 10. No abstract available. PMID 32791102
- [Derived] Gelb AF, Yamamoto A, Verbeken EK, Schein MJ, Moridzadeh R, Tran D, Fraser C, Barbers R, Elatre W, Koss MN, Glassy EF, Nadel JA. Further Studies of Unsuspected Emphysema in Nonsmoking Patients With Asthma With Persistent Expiratory Airflow Obstruction. Chest. 2018 Mar;153(3):618-629. doi: 10.1016/j.chest.2017.11.016. Epub 2017 Nov 29. PMID 29197547
- [Derived] Gelb AF, George SC, Camacho F, Fraser C, Flynn Taylor C, Shakkottai S. Increased nitric oxide concentrations in the small airway of older normal subjects. Chest. 2011 Feb;139(2):368-375. doi: 10.1378/chest.10-1157. Epub 2010 Aug 12. PMID 20705799
- [Derived] Gelb AF, George SC, Silkoff PE, Krishnan A, Fraser C, Taylor CF, Shinar CM, Maginot T. Central and peripheral airway/alveolar sites of exhaled nitric oxide in acute asthma. Thorax. 2010 Jul;65(7):619-25. doi: 10.1136/thx.2009.132696. PMID 20627920